CLINICAL TRIAL: NCT06243640
Title: Safety and Efficacy of Buagafuran Capsules in the Treatment of Generalized Anxiety Disorder: a Multi-center, Randomized, Double-blind, Double-dummy, Placebo-controlled, Positive-controlled, Fixed-dose Phase Ⅲ Clinical Trial
Brief Title: Phase 3 Clinical Trial of Buagafuran Capsules in the Treatment of GAD
Acronym: BGFN-2022-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Union Pharmaceutical Factory Ltd (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGFN-2022-02; 2022LB00288 (Registry Identifier: NMPA)
Record Dates: First submitted 2024-01-07; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — buagafuran; tebufenozide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose experimental group (Experimental): Subjects took 120mg per day of Buagafuran capsules after breakfast and dinner for 8 weeks
  Interventions: Drug: Buagafuran capsules, 15mg/ capsule
- Low-dose experimental group (Experimental): Subjects took 60mg per day of Buagafuran capsules and Buagafuran capsules mimic after breakfast and dinner for 8 weeks
  Interventions: Drug: Buagafuran capsules, 15mg/ capsule; Drug: Buagafuran capsules mimic, 0mg/ capsule
- Placebo-Control group (Placebo Comparator): Subjects took 0 mg per day Buagafuran capsules mimic after breakfast and dinner for 8 weeks
  Interventions: Drug: Buagafuran capsules mimic, 0mg/ capsule

INTERVENTIONS:
Drug: Buagafuran capsules, 15mg/ capsule — Subjects took Buagafuran capsules; twice per day, respectively, after breakfast and dinner for 8 weeks;
  Arms: High-dose experimental group; Low-dose experimental group
Drug: Buagafuran capsules mimic, 0mg/ capsule — Subjects took Buagafuran capsules mimic. twice per day, respectively, after breakfast and dinner for 8 weeks;
  Arms: Low-dose experimental group; Placebo-Control group

SUMMARY:
A placebo-controlled superiority design was used to evaluate the efficacy of 60 mg/ day or 120 mg/ day of Buagafuran capsules in the treatment of GAD

DETAILED DESCRIPTION:
This was a multi-center, randomized, double-blind, placebo-controlled, fixed-dose phase III clinical trial. Hierarchical factors for whether new generalized anxiety disorder (GAD) (new GAD vs. Non-new GAD).

Qualified subjects, according to the ratio of 1:1:1, were randomized into high-dose group, low-dose group and placebo-control group, and received a treatment course of 8 weeks. Participants were followed from baseline outpatient visit until end of the follow-up period( 10 weeks and 7 visits in total).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients aged 18-65 years old, of both sexes;
2. Met the diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for generalized anxiety disorder (GAD) and confirmed by the Brief International Neuropsychiatric Interview (M.I.N.I.);
3. The patient requires psychiatric medication;
4. Hamilton Anxiety Scale (HAMA) score ≥20, Hamilton Depression Scale (HAMD-17) score ≤2, Clinical Global Impression Scale (CGI-S) score ≥4 at screening and baseline Points;
5. Able to understand and voluntarily participate in this trial, signed informed consent.

Exclusion Criteria:

1. Patients with serious suicide risk at present, or HAMD-17 item 3-suicide score ≥3;
2. Patients with HAMD-17 > 17;
3. Patients whose HAMA scores decreased by ≥20% in the baseline period compared with the screening period:
4. Those who met the DSM-5 diagnostic criteria for other mental disorders except GAD;
5. Patients with previous history of depression, obsessive-compulsive disorder, bipolar disorder, psychotic disorder, factitious disorder and somatoform disorder; There were severe personality disorders, especially antisocial, borderline, or histrionic personality disorder, which were judged by the investigator to affect the patient's adherence to the study protocol;
6. Alcohol or drug abuse or dependence within 180 days before screening;
7. With severe or unstable has clinical significance of somatic disease, including any cardiovascular, cancer, kidney, respiratory, endocrine (including abnormal thyroid function), digestion, blood (such as with bleeding tendency) or nervous system diseases;
8. Patients whose physical examination or vital signs were abnormal and clinically significant (e.g. inadequately controlled hypertension, systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
9. Patients with a history of epilepsy or any other disease that may induce seizures, except convulsions caused by febrile convulsions in children;
10. Important abnormalities in laboratory tests during the screening period, such as abnormal liver function tests (alanine aminotransferase or aspartate transaminase > 2 times the normal value); Renal insufficiency (blood urea nitrogen or creatinine > 1.2 times the upper limit of normal);
11. Clinically significant abnormalities on electrocardiography (QT interval corrected by Fridericia method: ≥450 ms for men or ≥470 ms for women) or conditions deemed ineligible by the investigators;
12. Patients who had undergone psychiatric surgery, electroconvulsive therapy or transcranial magnetic stimulation within 90 days before screening;
13. Patients treated with β-blockers within 90 days before screening；
14. Patients with severe hypersensitivity, or allergic to at least 2 kinds of drugs (including photosensitivity);
15. Patients who had previously used two or more antidepressants and/or benzodiazepines at a clinically appropriate dose for at least 4 weeks but were still ineffective;
16. Receiving systemic psychotherapy or other non-pharmacological treatments (e.g., acupuncture, hypnosis, or phototherapy) within 6 weeks before the baseline visit;
17. Those who had used benzodiazepines within -7 to -1 days before screening, such as lorazepam, oxazepam, and alprazolam for less than 5 half-lives; The use of benzodiazepines with longer half-lives, such as diazepam, clonazepam, nitrazepam, estazolam, and flurazepam, not more than 5 half-lives or less than 30 days from the screening period, or the use of barbiturates not more than 5 half-lives or less than 30 days from the screening period;
18. Patients treated with monoamine oxidase inhibitors within -7 to 1 day before screening; Patients treated with fluoxetine within 30 days before screening;
19. Patients using antipsychotics, antidepressants and mood stabilizers with less than 5 half-lives before the baseline washout period;
20. Patients who discontinued traditional Chinese medicine, melatonin, and St. John's wort for less than 3 days before the baseline visit;
21. In the experimental drug delivery within 7 days before and during the test, cannot fast grapefruit or grapefruit juice;
22. Women during pregnancy or lactation experiments have fertility requirement (including men), and not to the male, the female patients is safe and effective contraceptive measures;
23. Unable to take medicine as prescribed;
24. Participants enrolled in other clinical trials within 90 days before screening;
25. Patients with other conditions deemed by the investigator to be ineligible for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton anxiety scale score after treatment | the end of week 8
  The Hamilton Anxiety (HAMA) Scale total score reflects the severity of the patients anxiety symptoms. The primary efficacy end point was the change from baseline to week 8 in HAMA total score to determine the superiority of buagafuran capsules over placebo. The larger the difference between buagafuran capsules over placebo, the better the curative effect.

SECONDARY OUTCOMES:
Change in each factor score and item score of Hamilton anxiety scale | the end of week 4 and 8
  One of the secondary efficacy end point was the change from baseline to week 4 and 8 in each factor score and item score of Hamilton anxiety scale to determine the superiority of buagafuran capsules over placebo. The larger the difference between buagafuran capsules over placebo, the better the curative effect.
Clinical global impression of improvement score | the end of week 4 and 8
  Subjective improvement of buagafuran capsules will be assessed using Clinical Global Impression of Improvement (CGI-I) score at week 4 and 8. The larger the difference between buagafuran capsules over placebo, the better the curative effect.
Clinical global impression of severity score | the end of week 4 and 8
  Subjective severity of buagafuran capsules will be assessed by the change from baseline to week 4 and 8 with Clinical global impression of severity (CGI-S) score, to determine the superiority of buagafuran capsules over placebo. The larger the difference between buagafuran capsules over placebo, the better the curative effect.
Complete remission rate | the end of week 8
  Complete remission rate was the proportion of subjects with HAMA total scale score ≤7 at the end of week 8. The larger the difference between buagafuran capsules over placebo, the better the curative effect.
Response rate | the end of week 8
  Response rate was the proportion of subjects with HAMA total score decreased by ≥50% from baseline to week 8. The larger the difference between buagafuran capsules over placebo, the better the curative effect.
Rapid-onset rate | the end of week 1 and 2
  Rapid-onset rate was the proportion of subjects with HAMA total score decreased by ≥20% from baseline to week 1 and 2. The larger the difference between buagafuran capsules over placebo, the better the curative effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Union Pharmaceutical Factory Ltd, Beijing, Beijing Municipality, China